CLINICAL TRIAL: NCT03258424
Title: A Phase I, Randomized, Placebo-Controlled, Study Designed to Assess the Safety, Tolerability, and Pharmacokinetics of PTI-428 in Subjects With Cystic Fibrosis.
Brief Title: Study Assessing PTI-428 Safety, Tolerability, and Pharmacokinetics in Subjects With Cystic Fibrosis on KALYDECO® as Background Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proteostasis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTI-428-05
Record Dates: First submitted 2017-08-18; First posted 2017-08-23 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PTI-428 (Active Comparator): Subjects will receive once daily dosing of PTI-428 or placebo for 14 days.
  Interventions: Drug: PTI-428
- Placebo (Placebo Comparator): Subjects will receive once daily dosing of PTI-428 or placebo for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTI-428 — PTI-428 or placebo will be given QD for 14 days.
  Arms: PTI-428
Drug: Placebo — PTI-428 or placebo will be given QD for 14 days.
  Arms: Placebo

SUMMARY:
The trial will consist of a single treatment group enrolling adult subjects with CF on background therapy with KALYDECO®. Approximately 16 subjects will be enrolled.

DETAILED DESCRIPTION:
The single treatment group will enroll adult subjects with CF currently on stable KALYDECO® background therapy for a minimum of 3 months at the time of randomization. Subjects will be randomized to either PTI-428 or placebo. Each dose will be administered once daily (QD) for a total of 14 Days. The subjects will continue treatment with KALYDECO® throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF.
* Stable on Kalydeco dosing for both label indication and per label dosing for a minimum of 3 months at the time of randomization
* Forced expiratory volume in 1 second (FEV1) 40-90% predicted.
* Non-smoker and non-tobacco user for a minimum of 30 days prior to screening and for the duration of the study.

Exclusion Criteria:

* Participation in another clinical trial or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer, prior to Study Day 1.
* History of cancer within the past five years (excluding cervical CIS with curative therapy for at least one year prior to screening and non-melanoma skin cancer).
* History of organ transplantation.
* Any sinopulmonary infection or CF exacerbation requiring a change or addition of medication (including antibiotics) within 1 month of Study Day 1 or any other clinically significant infection as determined by the investigator within 1 month of Day 1.
* History of alcohol or drug abuse or dependence within 12 months of screening as determined by the Investigator.
* Male and female of child-bearing potential, unless they are using highly effective methods of contraception during participation in the clinical study and for 4 weeks after termination from study.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by adverse events, safety labs, electrocardiograms (ECGs), physical examinations, and vital signs | Baseline through Day 21

SECONDARY OUTCOMES:
t1/2 of multiple oral doses | Baseline through Day 14
Tmax of multiple oral doses | Baseline through Day 14
Cmax of multiple oral doses | Baseline through Day 14
AUC0-t of multiple oral doses | Baseline through Day 14

OTHER OUTCOMES:
Change in nasal epithelial mRNA and protein expression over time | Baseline through Day 21
Change in sweat chloride over time | Baseline through Day 21
Change in FEV1 over time | Baseline through Day 21
Change in weight over time | Baseline through Day 21

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Celerion, Belfast
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: Yes